CLINICAL TRIAL: NCT00889031
Title: Protocol to Obtain Blood Samples for Leukemia Research
Status: Completed | Type: Observational
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Christopher H. Lowrey, Professor of Medicine and of Pharmacology and Toxicology, Dartmouth-Hitchcock Medical Center
Other Study IDs: D0905
Record Dates: First submitted 2009-04-24; First posted 2009-04-28 (Estimated); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: CLL
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 10cc of peripheral blood.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- No Treatment
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — Patients with Chronic Lymphocytic Leukemia (CLL)

SUMMARY:
The purpose of this study is to collect a blood sample in patients with Chronic Lymphocytic Leukemia (CLL).

DETAILED DESCRIPTION:
The blood sample will be used in the laboratory to perform studies focusing on Chronic Lymphocytic Leukemia (CLL).

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing routine blood draws as part of their ongoing follow-up for Chronic Lymphocytic Leukemia (CLL) at the Norris Cotton Cancer Center of DHMC.

Exclusion Criteria:

* Patients who have received cytotoxic drug, oral or intravenous steroid or targeted antibody therapy for CLL or other disease process within the past 6 months are excluded. Use of intravenous immunoglobulin (IVIg) is not a reason for exclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at Dartmouth-Hitchcock Medical Center's Norris Cotton Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 187 (Actual)
Dates: Start 2009-04 (Actual); Primary Completion 2018-03-09 (Actual); Study Completion 2018-03-09 (Actual)

PRIMARY OUTCOMES:
To determine the frequency with which CLL cells incubated ex vivo with vincristine undergo rapid interphase apoptosis. | 2 Years

SECONDARY OUTCOMES:
To determine whether suppression or inhibition of BCL2 family members can acutely sensitize CLL cells to vincristine. | 2 Years

CONTACTS AND LOCATIONS:
Overall Officials: Christopher H Lowrey, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

REFERENCES:
- [Background] Stadheim TA, Xiao H, Eastman A. Inhibition of extracellular signal-regulated kinase (ERK) mediates cell cycle phase independent apoptosis in vinblastine-treated ML-1 cells. Cancer Res. 2001 Feb 15;61(4):1533-40. PMID 11245462
- [Background] Vilpo JA, Koski T, Vilpo LM. Selective toxicity of vincristine against chronic lymphocytic leukemia cells in vitro. Eur J Haematol. 2000 Dec;65(6):370-8. doi: 10.1034/j.1600-0609.2000.065006370.x. PMID 11168494
- [Background] Kivekas I, Vilpo L, Vilpo J. Relationships of in vitro sensitivities tested with nine drugs and two types of irradiation in chronic lymphocytic leukemia. Leuk Res. 2002 Nov;26(11):1035-41. doi: 10.1016/s0145-2126(02)00050-4. PMID 12363473